CLINICAL TRIAL: NCT00244894
Title: Acupuncture for Hot Flashes in Prostate Cancer Patients
Brief Title: Acupuncture in Treating Hot Flashes in Patients With Prostate Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Tom Beer, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000445180; OHSU-7235; OHSU-HOR-02029-LX
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Fatigue; Hot Flashes; Prostate Cancer
Keywords: fatigue; recurrent prostate cancer; stage II prostate cancer; stage III prostate cancer; stage IV prostate cancer; hot flashes
MeSH Terms: conditions — Fatigue; Hot Flashes; Prostatic Neoplasms | interventions — Acupuncture Therapy; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: acupuncture therapy — Acupuncture treatments will be administered by a qualified practitioner twice a week for the first four weeks and once per week for an additional 6 weeks. Sterile, disposable Seirin needles will be placed bilaterally at the point Gallbladder 34, and along the spine at Bladder 15, Bladder 23, and Bladder 32. Low intensity electrostimulation at 2 Hz will be used for both Bladder 23 and Bladder 32. Points will also be placed unilaterally at Governing vessel 20, Heart 7, Pericardium 6, Liver 2, and Spleen 6
Procedure: fatigue assessment and management — Patients will utilize the Pittsburgh Sleep Quality Index (PSQI) to assess if the patient is an overall good sleeper or a poor sleeper.
Procedure: hot flashes attenuation — Patients will be asked to report hot flash frequency and severity daily using the hot flash diary (HFD) and hot flash severity guidelines (HFSG) throughout the treatment period.
Procedure: management of therapy complications — Short Form Health Survey (SF-36) will be used to assess the patient's overall vitality.
Procedure: quality-of-life assessment — Hot Flash Related Daily Interference Scale (HFRDIS)will be used to self-report hot flash related quality of life.

SUMMARY:
RATIONALE: Acupuncture may help relieve hot flashes in patients with prostate cancer.

PURPOSE: This clinical trial is studying how well acupuncture works in treating hot flashes in patients with prostate cancer who are undergoing androgen deprivation.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the impact of acupuncture therapy on the frequency and intensity of hot flashes and the quality of life of patients with prostate cancer undergoing androgen deprivation.
* Determine if blood serotonin and urinary 5-HIAA are increased in patients treated with acupuncture.
* Determine if plasma calcitonin gene-related peptide and MHPG are reduced in patients with hot flashes due to androgen deprivation treated with acupuncture.
* Determine the ability of tongue diagnosis, a traditional Chinese clinical assessment method, to predict clinical and biological changes in these patients.
* Determine the effect of acupuncture on insomnia and loss of vitality caused by hot flashes in these patients.

OUTLINE: Patients undergo acupuncture for 30 minutes twice weekly for 4 weeks and then once weekly for an additional 6 weeks.

Quality of life is assessed at baseline, at weeks 2, 4, 6, and 10, and then at 6 weeks after completion of study treatment.

After completion of study treatment, patients are followed at 6 weeks.

PROJECTED ACCRUAL: A total of 25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Confirmed diagnosis of prostate cancer
* Hot flash score ≥ 4 per day
* Prior or concurrent treatment with 1 of the following :

  * Bilateral orchiectomy
  * Gonadotropin releasing-hormone (GnRH) agonist or antagonist therapy
  * Antiandrogen therapy

PATIENT CHARACTERISTICS:

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* No mental impairment

PRIOR CONCURRENT THERAPY:

Chemotherapy

* No concurrent chemotherapy

Endocrine therapy

* See Disease Characteristics
* More than 4 weeks since prior estrogen or progestational drugs

Surgery

* See Disease Characteristics
* No prior placement of a pacemaker or other implantable electrical device

Other

* More than 4 weeks since prior gabapentin
* No concurrent antidepressant drugs

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2002-09; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Reduced hot flash frequency and intensity as measured by hot flash score from hot flash diary at 4 weeks after initiation of study treatment | Weeks 4 after initiation of study treatment.
Reduced hot flash frequency and intensity as measured by hot flash score from hot flash diary at 10 weeks after initiation of study treatment | 10 Weeks after initiation of study treatment.
Reduced hot flash frequency and intensity as measured by hot flash score from hot flash diary at 16 weeks after initiation of study treatment | 16 Weeks after initiation of study treatment.

SECONDARY OUTCOMES:
Improved quality of life as measured by hot flash related-quality of life (HFR-QOL) and elements of short form health survey (SF-36) at 4 weeks after initiation of study treatment | 4 Weeks after initiation of study treatment.
Change in biomarkers at baseline after initiation of study treatment | Baseline after initiation of study treatment.
Improved quality of life as measured by hot flash related-quality of life (HFR-QOL) and elements of short form health survey (SF-36) at 10 weeks after initiation of study treatment | 10 weeks after initiation of study treatment.
Improved quality of life as measured by hot flash related-quality of life (HFR-QOL) and elements of short form health survey (SF-36) at 16 weeks after initiation of study treatment | 16 Weeks after intiation of study treatment.
Change in biomarkers at 4 weeks after initiation of study treatment | 4 Weeks after initiation of study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz M. Beer, MD, Principal Investigator — OHSU Knight Cancer Institute
Locations (2):
- United States (2):
  - OHSU Knight Cancer Institute, Portland, Oregon
  - Portland VA Medical Center, Portland, Oregon